CLINICAL TRIAL: NCT04212702
Title: The Landscape of ESR1 Mutations in Asian Estrogen Receptor-positive Metastatic Breast Cancer Patients Detected by Liquid Biopsy and Impact on Hormonal Therapy-based Treatments
Brief Title: ESR1 Mutations in Asian ER+ Metastatic Breast Cancer on Hormonal Therapy-based Treatments
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Other Study IDs: 201703138RIPD
Record Dates: First submitted 2019-12-25; First posted 2019-12-27 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Everolimus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Approximately 8 ml plasma sample will be prepared from 20 ml whole blood to be used for circulating cell free DNA (cfDNA) extraction using the QIAamp Circulating Nucleic Acid Kit (Qiagen, Hilden, Germany, Cat. No. 55114). DNA concentration will be determined by the Qubit fluorometer (Thermo Fisher Scientific, Wilmington, DE, USA) and DNA integrity will be analyzed using the capillary electrophoresis (AATI Fragment analyzer).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Hormonal therapy-based treatments — Hormonal therapy-based treatments, ex. HT single agent, HT plus other targeted therapy, HT plus everolimus, HT plus metronomic oral chemotherapy or oral chemotherapy only
  Other Names: HT single agent, HT plus other targeted therapy, HT plus everolimus, HT plus metronomic oral chemotherapy or oral chemotherapy only

SUMMARY:
The investigator propose a prospective study using blood samples (liquid biopsy) of estrogen receptor (ER)-positive metastatic breast cancer (MBC) patients to understand the prevalence of estrogen receptor 1 (ESR1) mutation variants and the correlation with hormonal therapy (HT)-based treatment resistance in Asian ER-positive/human epidermal growth receptor-2 (HER2)-negative MBC population.

DETAILED DESCRIPTION:
The investigator will use next-generation targeted sequencing covering the entire ESR1 ligand-binding domain (LBD) region to understand 1. the spectrum and prevalence of specific ESR1 mutation variants in Asian women, and 2. the preliminary correlation of Asian-specific prevalent ESR1 LBD mutation variants such as Y537C with treatment efficacy. For the second purpose, the investigator will specifically focus on patients with ESR1 Y537C mutation, while the results from patients with wild type ESR1 and patients with D538G or Y537S mutant will be severed as control for preliminary comparison.

ELIGIBILITY:
Inclusion Criteria:

* (1) Female patients who are ≥ 20 years old at the time of informed consent.
* (2) Have histologically confirmed ER positive (defined as ≥1%) and/ or progesterone receptor (PR) positive (defined as ≥1%) breast cancer.
* (3) Have histologically confirmed HER2-negative breast cancer as defined by immuno-histochemistry (IHC) ≤ 2+, and/or fluorescence in situ hybridization (FISH) negative.
* (4) Patients who fits either one of the following two criteria are eligible: I. Have radiological or objective evidence of inoperable locally advanced or metastatic breast cancer and are planned to be given HT single agent, HT plus other targeted therapy, HT plus everolimus (reimbursed by National Health Insurance), HT plus metronomic oral chemotherapy or oral chemotherapy only by the treating physician. II. Locally advanced but operable patients before the resection of the primary tumor.

Exclusion Criteria:

* (1) Patients not suitable for oral anti-cancer treatment as determined by the investigator.
* (2) Known hypersensitivity to mammilian target of rapamycin (mTOR) inhibitors, e.g. Sirolimus (rapamycin).
* (3) Patients with a known history of HIV seropositivity. Screening for HIV infection at baseline is not required.
* (4) Patients being treated with drugs recognized as being strong inhibitors or inducers of the isoenzyme CYP3A.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Asian ER positive/HER2 negative metastatic breast cancer
Sampling Method: Probability Sample
Enrollment: 123 (Actual)
Dates: Start 2017-05-22 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
The percentage of ESR1 LBD mutation variant | 12 months
  The percentage of each ESR1 LBD mutation variant in Asian ER-positive/HER2-negative MBC who had received at least one line of HT

SECONDARY OUTCOMES:
Progression-free Survival (PFS) | 12 months
  PFS of patients who are treated with everolimus plus HT with either ESR1 wild type or different Asian-specific prevalent ESR1 LBD mutation variants such as Y537C

CONTACTS AND LOCATIONS:
Overall Officials: Yen-Shen Lu, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (2):
- Taiwan (2):
  - National Taiwan University Hospital, Taipei
  - Tri-Service General Hospital, Taipei